CLINICAL TRIAL: NCT03166293
Title: Early Intensive Exercise to Improve Walking in Children With Spastic Diplegia From Encephalopathy of Prematurity
Brief Title: Early Intensive Exercise to Improve Walking in Children With Spastic Diplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00072587
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Spastic Diplegia
Keywords: Cerebral Palsy; Physical Therapy; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive 3 months of intervention or 3 months of observation. Participants in the observation group will be offered the intervention once the observation period is complete
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Group (Experimental): Children will participate in intensive leg training with a physical therapist 1 hour/day, 4 days/week for 12 weeks. Children will continue to receive standard physical therapy care. Children will be followed for one year from the time of enrollment in the study.
  Interventions: Behavioral: Intensive leg training with a physical therapist
- Delay Group (Experimental): Children will be monitored for 3 months with no intervention. Children will participate in intensive leg training with a physical therapist after the 3 month delay period. Training will be 1 hour/day, 4 days/week for 12 weeks. They will continue to receive standard care throughout. Children will be followed for one year from the time of enrollment in the study.
  Interventions: Behavioral: Intensive leg training with a physical therapist

INTERVENTIONS:
Behavioral: Intensive leg training with a physical therapist — Intensive, self initiated activities of the lower extremities including walking over ground or on a treadmill (with or without support), kicking, jumping, standing balance, climbing stairs and slopes and other leg activities. Small weights will be added to the ankle and foot to increase the intensity of the exercise. A physical therapist will supervise sessions.
  Other Names: Therapist training

SUMMARY:
This is a randomized controlled trial comparing 3 months of intensive leg exercise to standard physiotherapy care for the improvement of motor function in the legs in young children with spastic diplegia.

DETAILED DESCRIPTION:
Children born prematurely are at risk of brain injury that can result in cerebral palsy(CP), most often affecting the legs, called spastic diplegia. Current treatment is largely passive, including leg braces, repeated injection of a paralyzing agent (Botox) in muscles that are abnormally active, and surgery as deformities occur. Active, physical therapy for weak muscles is infrequent, occurring twice a month or less. Yet, recent work with mammals show that early brain injury can be alleviated by intensive exercise therapy, but only while the animal is very young. Building on the success with early, intensive therapy for children with perinatal (around birth) stroke, the investigators will apply intensive therapy for the legs in children with diplegia. Children (8 mo - 3 yr old) will be randomly assigned to start treatment immediately or delay treatment for 3 mo. The delay period controls for improvement without treatment. These children will also receive treatment after the delay period. The therapy will be guided by physical therapists, and similar to the project on perinatal stroke. Children who live beyond commuting distance from the centres will form a 3rd group, whose parents will be coached by therapists to train the child at home. This group will show whether parents can be as effective as a therapist. Finally, when all children turn 4 yr old, they will be compared to other 4-yr-old children with the same diagnosis, but no training, to determine if there are long term benefits. The investigators anticipate that like the children with perinatal stroke, early intensive exercise will improve mobility, facilitate earlier and better walking, and that the effects will be enduring.

ELIGIBILITY:
Inclusion Criteria:

* children aged 8 mo - 3 yr old
* Evidence of periventricular white matter injury on diagnostic imaging
* clinical evidence of spastic diplegia

Exclusion Criteria:

* born before gestational age of 25 weeks
* birth weight <1000g (to exclude confounds related to extreme prematurity and low birth weights)
* MRI evidence of diffuse injury to the cerebral or cerebellar cortex
* uncontrolled epilepsy or infantile spasms in the past 6 months (contraindication for TMS)
* cardiovascular or musculoskeletal complications that preclude participation in intensive exercise
* Botulinum toxin (BTX-A) injections in the last 6 months
* Predicted GMFCS 4 or 5

Ages: 8 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Functional Measure - 66 Items (GMFM-66) over 3 months | Baseline, 3 months
  This is a 66 item criterion-referenced observational measure to assess change in gross motor function of children with cerebral palsy.

SECONDARY OUTCOMES:
Change in forces during treadmill walking over 3 months | Baseline, 3 months
  The child will be supported to walk on a treadmill while we record the leg motions and the forces under the feet during walking.

CONTACTS AND LOCATIONS:
Overall Officials: Jaynie Yang, PhD, Principal Investigator — University of Alberta; Monica Gorassini, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No